CLINICAL TRIAL: NCT06444828
Title: Outcome Following Reverse Shoulder Arthroplasty for Acute Proximal Humerus Fractures in Patients 60 Years of Age and Older With Different Inclination Implants Versus Non-surgical Treatment- Trial Protocol: a Prospective RCT, Single Blinded
Brief Title: Comparing Outcomes of Non-surgical Versus Surgical Treatment of Shoulder Fractures With Different Shoulder Replacements
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Southern Denmark (Other)
Collaborators: Region of Southern Denmark (Other)
Responsible Party: Principal Investigator, Klaus Wilhelm Josef Hanisch, Principal Investigator, University of Southern Denmark
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ISRCTN85422168
Record Dates: First submitted 2023-11-30; First posted 2024-06-06 (Actual); Last update posted 2024-12-11 (Actual); Status verified 2024-12

CONDITIONS: Proximal Humeral Fracture; Humeral Head Fracture
Keywords: proximal humerus fracture; Reverse Shoulder Arthroplasty
MeSH Terms: conditions — Shoulder Fractures

STUDY DESIGN:
Intervention Model Description: RCT, single blinded
Who Masked: Participant
Masking Description: non information of the type of implant used is given to the patient
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- non operative treatment (No Intervention): Proximal humeral fractures (PHF) treated non-operative, Rehabilitation only
- Reverse Shoulder Arthroplasty (RSA) (Active Comparator): RSA 135/ 155 inclination
  Interventions: Procedure: Non-operative

INTERVENTIONS:
Procedure: Non-operative — Non-operative treatment versus operative treatment (surgery)
  Other Names: Surgery Reverse Shoulder Arthroplasty
  Arms: Reverse Shoulder Arthroplasty (RSA)

SUMMARY:
The optimal treatment of complex shoulder fracture is controversial. In general, non-surgical treatment is recommended for older patients, but results are often unsatisfying. Therefore different surgical approaches have been tried to improve outcomes for this group of patients. Reverse shoulder arthroplasty has shown promising results for these types of fractures and changes in the design of the implant might improve outcomes further. The aim of this study is to compare the outcomes of complex shoulder fractures after non-surgical versus surgical treatment and compare two different types of implants.

DETAILED DESCRIPTION:
The optimal treatment of proximal humeral fracture (PHF) Neer type III and IV AO B1.1,1.2 and C1.1,3.1 is controversial. National guidelines for Denmark have been published in 2015 and updated 2019. They recommend conservative treatment to all kinds of PHF for patients aged above 60 years. Exceptions are fracture-dislocations, headsplits or surgical conditions, where intervention is mandatory like open fractures and impaired nerve- and circulation.

Recently reverse shoulder arthroplasty (RSA) has gained expanding popularity in treating PHF . Compared with osteosynthesis (ORIF) or hemiarthroplasty (HA) outcomes were superior , . The importance of tuberosity healing for good functional outcomes has lead to development of different implants and fixation techniques. The original RSA design by Grammont with 155 degree inclination of the humeral stem was made for cuff-arthropathy. This design moves the center of rotation in a medial direction, and increase the tension on the tuberosities.

In contrast "anatomical" designed humeral implants with 135 degree enables more anatomical refixation of the tuberosities with less tension and might reduce the risk of resorption or displacement of the fragments. To implant a 155 degree RSA the surgeon has to remove parts of the rotator cuff, to enable the sliding rotation. On the other hand with a 135 degree inclination humeral component, a cuff sparing technique is possible.

The aim of this study is to compare outcomes of two different designed RSA stems versus conservative treatment of PHF Neer type III or IV / AO B&C.

ELIGIBILITY:
Inclusion Criteria:

Displaced Proximal Humeral Fractures (PHF) Neer type III or IV / AO B&C. Radiological confirmed

Exclusion Criteria:

other types of PHF, Head splits, gleno-humeral dislocations, pathological fractures. Refuse to participate in the study. Non-compliant, drug/alcohol abuse or institutionalized, (Low-cooperative),

Ages: 60 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2021-09-01 (Actual); Primary Completion 2025-09-01 (Estimated); Study Completion 2026-09-01 (Estimated)

PRIMARY OUTCOMES:
The primary outcome is Western Ontario Osteoarthritis of the Shoulder Index (WOOS) | one years follow up (FU)
  All participants are assessed with online questionnaire, Patient Related Outcome Measurement (PROM) 0-100% (100% best), validated

SECONDARY OUTCOMES:
Constant Murley score | one and two years FU
  All participants are assessed with function scores. 0-100% (100% best) by physiotherapist
Subjective shoulder Volume (SSV) | one and two years FU
  All participants are assessed with online questionnaire PROM 0-100% (100% best)
x-rays | one and two years FU
  stating healing, displacement, resorbtion of the tuberosities

CONTACTS AND LOCATIONS:
Overall Officials: Klaus Hanisch, Study Chair — University of Southern Denmark
Locations (1):
- University Hospital Southern Danmark, Esbjerg, South, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: ISRCTN — http://doi.org/10.1186/ISRCTN85422168

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-06-06): https://cdn.clinicaltrials.gov/large-docs/28/NCT06444828/Prot_SAP_000.pdf